CLINICAL TRIAL: NCT03900637
Title: Multi-institutional Study to Increase Breast Conserving Surgery (BCS) Rate With Personalized Neoadjuvant Strategy in ER Positive and HER2 Negative Breast Cancer Patients for Whom BCS is Not Feasible
Brief Title: PersonaLized neoAdjuvant Strategy ER Positive and HER2 Negative Breast Cancer TO Increase BCS Rate
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonshik Han, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLATO study
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Leuprolide; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): 1. MammaPrint high risk :
     * Neoadjuvant chemotherapy : Adriamycin/Cyclophosphamide #4 followed by Docetaxel #4
  2. MammaPrint low risk :
     * Premenopausal women : Letrozole 2.5mg PO QD + leuprorelin acetate 3.6mg SQ every 4weeks during 16 weeks (if needed, maximum for 24 weeks)
     * Postmenopausal women : Letrozole 2.5mg PO QD during 16 weeks (if needed, maximum for 24 weeks)
  Interventions: Drug: Leuprorelin acetate; Drug: Letrozole; Genetic: MammaPrint

INTERVENTIONS:
Drug: Leuprorelin acetate — In premenopausal women, 3.75mg of leuprorelin acetate is subcutaneously administered once every 4 weeks for 16 weeks. (if needed, maximum for 24 weeks)
  Other Names: Leuplin
Drug: Letrozole — 2.5 mg tablet is orally administered once a day, without regard to meals, for 16 weeks (if needed, maximum for 24 weeks)
  Other Names: Lenara; Bretra
Genetic: MammaPrint — In this study, patients with MammaPrint test is performed, neoadjuvant chemotherapy is conducted to genomic High Risk patients, and neoadjuvant endocrine therapy is conducted to Low Risk patients.

SUMMARY:
In ER+ and HER2- breast cancer(BC) patients for whom BCS is not feasible, we investigate the rate of BCS can be increased while decreasing unnecessary chemotherapy thru selective neoadjuvant chemotherapy or neoadjuvant endocrine therapy using tools of nodal status, Ki-67, and multigene assay(Mammaprint)

DETAILED DESCRIPTION:
In patients with resectable BC, the neoadjuvant chemotherapy is recognized as one of the standard therapy in order to control and prevent the micrometastasis.

Conducting neoadjuvant chemotherapy can lead to increased numbers of BCS compared with adjuvant chemotherapy and the prognosis of BC patients is known to be improved when there is pathological complete response (pCR) after neoadjuvant chemotherapy compared with no pCR.

The effect of neoadjuvant chemotherapy is different in breast cancer subtypes. The quasi-pCR in HR- HER2+ BC is reported as 67% while 37% and 13% in triple negative and HR+ HER2- BC, respectively and it indicates that neoadjuvant chemotherapy has only limited effect in HR+ BC and the declined quality of life and the fecundity loss due to chemotherapy is a serious socioeconomic loss, especially in young patients.

According to the SOFT trial, for high risk, pre-menopausal women, use of exmestane (AI, Aromatase Inhibitors) and ovarian suppression as adjuvant systemic therapy did improve the PFD compared with the use of tamoxifen and ovarian suppression.

Neoadjuvant hormonal therapy as well as neoadjuvant chemotherapy has benefits in making inoperable BC to operable BC and improving the possibility of BCS by reducing the tumor size with complete response or partial response. Although these neoadjuvant systemic therapies have an ultimate objective to reduce the recurrence rate and improve the survival rate, the overall survival and disease-free survival has been reported similar to adjuvant systemic therapies. The clinical response rate of neoadjuvant hormonal therapy ranged from 13.5% to 100%, the radiologic response rate by ultrasound ranged from 20% to 91.7%, and these are statistically similar to the response rate of the neoadjuvant chemotherapy in ER+ patients. Most studies where letrozole was tested among AIs showed that letrozole has a similar or a little better effect on clinical or radiological response rate over tamoxifen and there were statistically more patients who became operable or eligible for BCS after neoadjuvant chemotherapy. Comparison studies among AIs showed that the response rates have been best achieved in letrozole over anastrozole and exemestane and the BCS rate was lowest in letrozole without statistical significance. According to the standard treatment guideline suggesting the selective use of ovarian suppression along with tamoxifen in HR+, premenopausal patients, a study investigated the combined treatment of letrozole with reversible ovarian ablation using goserelin (luteinizing hormone-releasing hormone: LHRH). The results showed that the response rate of the combination treatment of goserelin and anastrozole for 24 weeks as neoadjuvant hormonal therapy was statistically superior to goserelin and tamoxifen in premenopausal BC patients and this was not observed in the adjuvant setting. The most commonly used agents in BC are goserelin and leuprorelin(Leuplin) and their mechanism of action is to desensitize the hypothalamus and suppress the ovarian function by reducing the secretion of LH and FSH.

MammaPrint, which analyses 70-gene expressed in breast cancer, can identify low risk patients who may safely forgo chemotherapy and high risk patients who can benefit from chemotherapy. Recent results from MINDACT trial have proved that 46.2% of HR+ and clinical high risk patients were classified into MammaPrint low risk and they could avoid unnecessary chemotherapy. In 2017 San Antonio breast cancer symposium, Dubsky et al. reported the analysis of correlation between neoadjuvant chemotherapy and score of Endopredict(EP) multigene assay in ER+ and HER2- patients treated on ABCSG 34. In neoadjuvant chemotherapy group, reduction of tumor size in patients with low EP score(Endopredict low risk group) was significantly low(NPV 100%). Meanwhile, in neoadjuvant hormonal therapy group, reduction of tumor size in patients with high EP score(Endopredict high risk group) was significantly low(NPV 92%). These results support the evidence that response of neoadjuvant chemotherapy or hormonal therapy can be predicted by the molecular score of tumor and selective treatment can maximize the effect.

Accordingly, in this study, patients with MammaPrint test is performed, neoadjuvant chemotherapy is conducted to genomic High Risk patients, and neoadjuvant endocrine therapy is conducted to Low Risk patients. Although adjuvant therapy is conducted after the completion of this study, in case there is progressive disease (PD) after neoadjuvant endocrine therapy, adjuvant chemotherapy is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically and immunohistochemically confirmed ER+ and HER2- BC patients
2. Stage I-IIIA BC patients with detectable tumor sizes
3. BC patients for whom BCS is not feasible due to tumor sizes or locations (two surgeons at each institution evaluate the infeasibility of BCS)
4. Patients without distant metastasis which were identified pathologically or radiologically
5. Female patients ≥ 19 years

   * Diagnosis of menopause is defined as no menstruation for 1-year or both ovaries removed surgically
6. ECOG 0-2
7. Patients with adequate bone marrow function

   * Hemoglobin 10 g/dL, ANC 1,500/mm3, Plt 100,000/mm3
8. Patients with adequate kidney function

   * serum Cr ≤ 1.5 mg/dL
9. Patients with adequate liver function

   * Bilirubin: ≤ 1.5 times of upper normal limit
   * AST/ALT: ≤ 1.5 times of upper normal limit
   * Alkaline phosphatase: ≤ 1.5 times of upper normal limit
10. Patients who decided to voluntarily participate in this trial with written informed consent

Exclusion Criteria:

1. History of treatment for ipsilateral BC or breast carcinoma in situ
2. Confirmed distant metastasis of BC
3. History of cancer other than BC
4. Pregnant (positive pregnancy test within a week of enrollment) or breast-feeding patients
5. Uncontrolled severe infection
6. Psychiatric illness or epilepsy
7. Male BC patients
8. Inability to understand and willingness to sign a written informed consent
9. Mammographic extensive microcalcification
10. Multicentral, Bilateral BC
11. History of chemotherapy or endocrine therapy on contralateral BC for the past 2 years
12. ER-
13. HER2+
14. Undetectable and unmeasurable primary tumor size

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion Rate | 4 months(maximum 6 months)
  Evaluate the conversion rate from BCS-ineligible to BCS-eligible patients

SECONDARY OUTCOMES:
Actual Conversion Rate | 4 months(maximum 6 months)
  Evaluate the actual performance rate of BCS
pCR | 4 months(maximum 6 months)
  Evaluate pathological complete response
cCR | 4 months(maximum 6 months)
  Evaluate clinical response rate
Tumor Size Reduction Rate | 4 months(maximum 6 months)
  Evaluate the accomplished rate of targeted tumor size reduction which enable to make BCS possible at presentation

OTHER OUTCOMES:
DFS | 5 years
  Evaluate disease free survivals
IBTR | 5 years
  Evaluate ipsilateral breast tumor recurrence
Blueprint subtype | 4 months(maximum 6 months)
  Evaluate response rate by Blueprint subtype

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea